CLINICAL TRIAL: NCT03996928
Title: Eccentric Exercise in Epicondylitis: Direct Application By Physical Therapist Vs Self-Application By Patient
Brief Title: Eccentric Exercise in Epicondylitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Andaluz Health Service (Other Government)
Responsible Party: Principal Investigator, ANTONIO OYA CASERO, Principal Investigator, Andaluz Health Service
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OYA-EXC-2019-1
Record Dates: First submitted 2019-06-22; First posted 2019-06-25 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Tendinopathy
Keywords: Epicondylitis; Tennis elbow; Eccentric exercise
MeSH Terms: conditions — Tendinopathy; Tennis Elbow | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Single blind randomized controlled trial
  INDEPENDENT VARIABLES
  Age, Sex, Work activity (referred to a superior member): intense -including, among other kind of activities, keyboards users and housewives-light.
  Basal pain according to visual analogue scale (VAS) of 100 mm. Baseline disability according to the DASH questionnaire (Disabilities of the Arm, Shoulder and Hand), which is self-administered.
  DEPENDENT VARIABLES
  Pain according to the aforementioned scale just after treatment (2 weeks) and at 3 months.
  Disability according to the aforementioned questionnaire just after the treatment (2 weeks) and at three months.
  Satisfaction with the treatment right after it (2 weeks) and at three months. A Likert scale of five points ( very satisfied, satisfied, neither satisfied nor unsatisfied, very unsatisfied) will be used.
  Co-interventions (Systemic and/or topical route drugs, physiotherapy modalities received outside the system, use of orthoses).
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eccentric exercise by physiotherapist (Experimental): A physiotherapist will apply (in this order) a plan of stretching exercises, warm-up exercises and eccentric exercises of epicondylar muscle,according to a program of 10 sessions of 20 minutes each, during two weeks.
  Before exercise, ultrasounds will be applied at intensity of 0.1 wat/cm2, which is considered as a placebo, in order to achieve greater adherence and monitor the treatment.
  Interventions: Other: Exercise
- Illustrated booklet (Active Comparator): A physiotherapist will train the patient an exercise plan equivalent to the one above explained with the help of illustrations. Now, in order to achieve palmar flexion at the same time the patients will contract their epicondylar muscles (the eccentric effect), and elastic band is used.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise

SUMMARY:
There is more and more evidence of the importance of the role of kinesitherapy in the management of epicondylitis, specifically (but not exclusively) of eccentric exercise. Since eccentric kinesitherapy, when applied in a systematic way by a physiotherapist, consumes time and human resources in a significant way, and in the case of such a prevalent pathology, it is frequent that strategies of training the patient are addressed so that this is who perform the exercises after learning them. However, it is not proven that the efficacy and safety of this approach is equivalent to treatment applied by a physiotherapist.

A randomized single-blind controlled trial is conducted that compares both treatment approaches for epicondylitis (eccentric exercises applied directly by a physiotherapist for 10 sessions, and eccentric exercises applied by the patient during the same time) in terms of efficacy against pain, functionality and patient satisfaction, all this within the framework of the public health system.

DETAILED DESCRIPTION:
The main objective of this study is:

To compare the efficacy of an eccentric exercise program applied to patients with epicondylosis by a structured manual program in ten sessions and by an illustrated booklet.

The specific objectives of this study are:

Compare the effectiveness of the above-cited approaches in terms of pain Compare the effectiveness of the above-cited approaches in terms of function Compare the effectiveness of the above-cited approaches in terms of satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years old
* Epicondylosis of three or more months of evolution.
* Acceptance of the voluntary participation in the study and signature of the informed consent.

Exclusion Criteria:

* Generalized musculoskeletal pain.
* Rheumatological affections involving of the upper limb.
* Cervicobrachialgia.
* Previous trauma in upper limb.
* Neurological or other pathology that may interfere with the function of the upper limb.
* Being out of work or in litigation due to the pathology of the upper limb.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale of pain | At two weeks
  The Visual Analogue Scale (VAS) quantifies of pain described by the patient with maximum reproducibility among observers. It consists of a 10-centimeter horizontal line, at the ends of which the extreme expressions of a symptom are marked: no pain on the left wiht a score 0, and the highest possible pain on the right wiht a score 10. The patient is asked to mark the point that indicates the intensity in the line and is measured with a millimeter ruler. The intensity is expressed in centimeters or millimeters.
  A value lower than 4 in the VAS means mild or mild-moderate pain, a value between 4 and 6 implies the presence of moderate-severe pain, and a value greater than 6 implies the presence of very intense pain.
Visual analogue scale of pain | Three months
  The Visual Analogue Scale (VAS) quantifies of pain described by the patient with maximum reproducibility among observers. It consists of a 10-centimeter horizontal line, at the ends of which the extreme expressions of a symptom are marked: no pain on the left wiht a score 0, and the highest possible pain on the right wiht a score 10. The patient is asked to mark the point that indicates the intensity in the line and is measured with a millimeter ruler. The intensity is expressed in centimeters or millimeters.
  A value lower than 4 in the VAS means mild or mild-moderate pain, a value between 4 and 6 implies the presence of moderate-severe pain, and a value greater than 6 implies the presence of very intense pain.
Quick-Dash | At two weeks
  At least 10 of the 11 questions must be completed to calculate the score Disability / Symptom of Quick DASH.
  The assigned values for all the complete answers are summed and averaged, giving as a result, a score based on five. This value is then taken to a score based on 100 subtracting 1 and multiplying it by 25. A higher score greater disability.
Quick-Dash | Three months
  At least 10 of the 11 questions must be completed to calculate the score Disability / Symptom of Quick DASH.
  The assigned values for all the complete answers are summed and averaged, giving as a result, a score based on five. This value is then taken to a score based on 100 subtracting 1 and multiplying it by 25. A higher score greater disability.
Satisfaction questionnaire | At two weeks
  A survey will be carried out to find out what the patient has perceived by asking a question about his satisfaction with the treatment received, choosing one of the following answers:
  1. Very satisfied
  2. Satisfied
  3. Neither satisfied nor unsatisfied
  4. Unsatisfied
  5. Very unsatisfied
Satisfaction questionnaire | Three months
  A survey will be carried out to find out what the patient has perceived by asking a question about his satisfaction with the treatment received, choosing one of the following answers:
  1. Very satisfied
  2. Satisfied
  3. Neither satisfied nor unsatisfied
  4. Unsatisfied
  5. Very unsatisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Antonio Oya Casero, Jaén, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weber C, Thai V, Neuheuser K, Groover K, Christ O. Efficacy of physical therapy for the treatment of lateral epicondylitis: a meta-analysis. BMC Musculoskelet Disord. 2015 Aug 25;16:223. doi: 10.1186/s12891-015-0665-4. PMID 26303397
- [Background] Abate M, Silbernagel KG, Siljeholm C, Di Iorio A, De Amicis D, Salini V, Werner S, Paganelli R. Pathogenesis of tendinopathies: inflammation or degeneration? Arthritis Res Ther. 2009;11(3):235. doi: 10.1186/ar2723. Epub 2009 Jun 30. PMID 19591655
- [Background] Nagrale AV, Herd CR, Ganvir S, Ramteke G. Cyriax physiotherapy versus phonophoresis with supervised exercise in subjects with lateral epicondylalgia: a randomized clinical trial. J Man Manip Ther. 2009;17(3):171-8. doi: 10.1179/jmt.2009.17.3.171. PMID 20046624
- [Background] Murgia A, Harwin W, Prakoonwit S, Brownlow H. Preliminary observations on the presence of sustained tendon strain and eccentric contractions of the wrist extensors during a common manual task: implications for lateral epicondylitis. Med Eng Phys. 2011 Jul;33(6):793-7. doi: 10.1016/j.medengphy.2011.02.002. Epub 2011 Mar 16. PMID 21414830
- [Background] Gautam VK, Verma S, Batra S, Bhatnagar N, Arora S. Platelet-rich plasma versus corticosteroid injection for recalcitrant lateral epicondylitis: clinical and ultrasonographic evaluation. J Orthop Surg (Hong Kong). 2015 Apr;23(1):1-5. doi: 10.1177/230949901502300101. PMID 25920633
- [Background] Jindal N, Gaury Y, Banshiwal RC, Lamoria R, Bachhal V. Comparison of short term results of single injection of autologous blood and steroid injection in tennis elbow: a prospective study. J Orthop Surg Res. 2013 Apr 27;8:10. doi: 10.1186/1749-799X-8-10. PMID 23621906
- [Background] Johnson GW, Cadwallader K, Scheffel SB, Epperly TD. Treatment of lateral epicondylitis. Am Fam Physician. 2007 Sep 15;76(6):843-8. PMID 17910298
- [Background] Viola L. A critical review of the current conservative therapies for tennis elbow (lateral epicondylitis). Australas Chiropr Osteopathy. 1998 Jul;7(2):53-67. PMID 17987156
- [Background] Bisset LM, Collins NJ, Offord SS. Immediate effects of 2 types of braces on pain and grip strength in people with lateral epicondylalgia: a randomized controlled trial. J Orthop Sports Phys Ther. 2014 Feb;44(2):120-8. doi: 10.2519/jospt.2014.4744. Epub 2014 Jan 9. PMID 24405258
- [Background] Speed C. A systematic review of shockwave therapies in soft tissue conditions: focusing on the evidence. Br J Sports Med. 2014 Nov;48(21):1538-42. doi: 10.1136/bjsports-2012-091961. Epub 2013 Aug 5. PMID 23918444
- [Background] Olaussen M, Holmedal O, Mdala I, Brage S, Lindbaek M. Corticosteroid or placebo injection combined with deep transverse friction massage, Mills manipulation, stretching and eccentric exercise for acute lateral epicondylitis: a randomised, controlled trial. BMC Musculoskelet Disord. 2015 May 20;16:122. doi: 10.1186/s12891-015-0582-6. PMID 25989985
- [Background] Cullinane FL, Boocock MG, Trevelyan FC. Is eccentric exercise an effective treatment for lateral epicondylitis? A systematic review. Clin Rehabil. 2014 Jan;28(1):3-19. doi: 10.1177/0269215513491974. Epub 2013 Jul 23. PMID 23881334
- [Background] Raman J, MacDermid JC, Grewal R. Effectiveness of different methods of resistance exercises in lateral epicondylosis--a systematic review. J Hand Ther. 2012 Jan-Mar;25(1):5-25; quiz 26. doi: 10.1016/j.jht.2011.09.001. Epub 2011 Nov 9. PMID 22075055
- [Background] Peterson M, Butler S, Eriksson M, Svardsudd K. A randomized controlled trial of eccentric vs. concentric graded exercise in chronic tennis elbow (lateral elbow tendinopathy). Clin Rehabil. 2014 Sep;28(9):862-72. doi: 10.1177/0269215514527595. Epub 2014 Mar 14. PMID 24634444
- [Background] Soderberg J, Grooten WJ, Ang BO. Effects of eccentric training on hand strength in subjects with lateral epicondylalgia: a randomized-controlled trial. Scand J Med Sci Sports. 2012 Dec;22(6):797-803. doi: 10.1111/j.1600-0838.2011.01317.x. Epub 2011 Apr 18. PMID 21496112
- [Background] Tyler TF, Thomas GC, Nicholas SJ, McHugh MP. Addition of isolated wrist extensor eccentric exercise to standard treatment for chronic lateral epicondylosis: a prospective randomized trial. J Shoulder Elbow Surg. 2010 Sep;19(6):917-22. doi: 10.1016/j.jse.2010.04.041. Epub 2010 Jun 26. PMID 20579907
- [Background] Burge E, Monnin D, Berchtold A, Allet L. Cost-Effectiveness of Physical Therapy Only and of Usual Care for Various Health Conditions: Systematic Review. Phys Ther. 2016 Jun;96(6):774-86. doi: 10.2522/ptj.20140333. Epub 2015 Dec 17. PMID 26678447
- [Background] Korthals-de Bos IB, Smidt N, van Tulder MW, Rutten-van Molken MP, Ader HJ, van der Windt DA, Assendelft WJ, Bouter LM. Cost effectiveness of interventions for lateral epicondylitis: results from a randomised controlled trial in primary care. Pharmacoeconomics. 2004;22(3):185-95. doi: 10.2165/00019053-200422030-00004. PMID 14871165